CLINICAL TRIAL: NCT05142137
Title: Randomised, Placebo-controlled Chronic Study to Investigate Gastrointestinal Tolerability of a Novel Alpha Glucan in Adults
Brief Title: Novel Alpha Glucan GI Tolerability Study (Loris Chronic)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Société des Produits Nestlé (SPN) (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 2025NR
Record Dates: First submitted 2021-09-02; First posted 2021-12-02 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2021-11

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Intervention Model Description: 3x3
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Novel alpha glucan_dose1 (Experimental): Total of 180 g of the novel alpha glucan per day, consumed in 4 individual doses (i.e. 4x45 g, with each dose dissolved in 300 ml of water)
  Interventions: Dietary Supplement: Drinkable solution
- Novel alpha glucan_dose2 (Experimental): Total of 80 g of the novel alpha glucan + 100 g glucose syrup per day, consumed in 4 individual doses (i.e. 4x45 g, with each dose dissolved in 300 ml of water)
  Interventions: Dietary Supplement: Drinkable solution
- glucose syrup (Active Comparator): Total of 180 g glucose syrup per day, consumed in 4 individual doses (i.e. 4x45 g, with each dose dissolved in 300 ml of water).
  Interventions: Dietary Supplement: Drinkable solution

INTERVENTIONS:
Dietary Supplement: Drinkable solution — The volunteers will consume 300 ml of liquid solution containing the novel alpha glucan or glucose syrup

SUMMARY:
This study aims to evaluate the gastrointestinal tolerance of chronic consumption (7 days) of a novel alpha glucan compared to a rapidly available carbohydrate (glucose syrup).

DETAILED DESCRIPTION:
This study will be randomized, double blind, placebo-controlled, single-center, and 3x3 crossover in design.

Eligible participants will be randomized to receive the below products in single dose and in different random sequence, as determined by the randomization system:

1. novel alpha glucan (80 g/day)
2. novel alpha glucan (180 g/day)
3. glucose syrup (180 g/day)

ELIGIBILITY:
Inclusion Criteria:

1. Male or female participant,
2. Healthy status (based on anamnesis),
3. Age between 18 and 65 years,
4. Body mass index (BMI) between 18.5 and 29.9 kg/m2,
5. Able to understand and sign informed consent form,
6. Having a smartphone with Android or iOS version compatible with Patient Cloud application

Exclusion Criteria:

1. Fasting plasma glucose higher or equal to 6,1 mmol /L at screening,
2. Type I and type 2 diabetes,
3. Pregnant or lactating women,
4. Known food allergy or intolerance to test products,
5. Treatment with anorectic drugs, glucose-lowering drugs, steroids, medications known to affect glucose metabolism and/or gastric motility, or any condition known to affect gastro-intestinal integrity and food absorption,
6. Colonoscopy, irrigoscopy or other bowel cleansing procedures four weeks prior the test,
7. Any concomitant medication potentially interfering with study procedures and assessment: such as antibiotics, antiacids, or other medications impacting transit time,
8. Major medical/surgical event in the last 3 months potentially interfering with study procedures and assessments,
9. Abnormal bowel transit, history of a gastrointestinal disorder (e.g., inflammatory bowel disease, diverticular diseases, colon cancer), or history of chronic constipation with passage of fewer than 3 spontaneous bowel movements per week on average or chronic or recurrent diarrhea with spontaneous bowel movements more often than 3 times daily,
10. Recent episode of an acute gastrointestinal illness,
11. Habitual consumption of more than four servings per day of high-fiber foods or extreme dietary habits (e.g. very low carbohydrate diet),
12. Ongoing or recent weight loss interventions (e.g. dietary weight loss programs),
13. Alcohol intake higher than 2 servings per day. A serving is 0.4 dl of strong alcohols, 1 dl of red or white wine, or 3 dl of beer,
14. Score of "severe" symptom for any of the symptoms included in the gastrointestinal symptom questionnaire,
15. Volunteer who cannot be expected to comply with the protocol,
16. Family or hierarchical relationships with Clinical Innovation Lab team.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2021-08-16 (Actual); Primary Completion 2021-10-11 (Actual); Study Completion 2021-10-31 (Actual)

PRIMARY OUTCOMES:
Gastrointestinal Symptom Rating Scale (GSRS) | Throughout 7 days of treatment
  Validated questionnaire exploring the presence and severity of GI symptoms over the previous 7 days. The GSRS is a disease-specific instrument of 15 items combined into five symptom clusters depicting reflux, abdominal pain, indigestion, diarrhea and constipation. The GSRS has a seven-point graded Likert-type scale where 1 represents absence of troublesome symptoms and 7 represents very troublesome symptoms. The effect of the interventions on the GSRS will be assessed by a linear mixed model and will take into account information on this from all 7 days of treatment.

SECONDARY OUTCOMES:
Stool consistency | Throughout 7 days of treatment
  The Bristol stool scale is a diagnostic medical tool designed to classify the form of human faeces into seven categories. Types 1 and 2 indicate constipation, with 3 and 4 being the ideal stools, whereas 5 indicate lack of dietary fiber, and 6 and 7 indicate diarrhoea. The effect of the interventions on stool consistency will be assessed by a linear mixed model and will take into account information on this from all 7 days of treatment.
Stool frequency | Throughout 7 days of treatment
  The participants report the number of defecations they have per day, throughout the 7 days study period. There is a large variability in this, but typically 1-3 defecations per day is considered normal, whereas more indicate a runny stool, and fewer a tendency for constipation. The effect of the interventions on stool frequency will be assessed by changes in stool frequency over time, taking all information on this from all 7 days of treatment into account.

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Innovation Lab, Lausanne, Canton of Vaud, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kelly RM, Dijkhuizen L, Leemhuis H. Starch and alpha-glucan acting enzymes, modulating their properties by directed evolution. J Biotechnol. 2009 Mar 25;140(3-4):184-93. doi: 10.1016/j.jbiotec.2009.01.020. Epub 2009 Feb 7. PMID 19428713
- [Background] Synytsya A, Novak M. Structural analysis of glucans. Ann Transl Med. 2014 Feb;2(2):17. doi: 10.3978/j.issn.2305-5839.2014.02.07. PMID 25332993